CLINICAL TRIAL: NCT03878511
Title: Effect of Vaginal Lactose on the Vaginal Microbiota in Women With Bacterial Vaginosis: Double-blind, Placebo-controlled Randomised Trial
Brief Title: Therapeutic Lactose to Support Vaginal Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Humaidan (Other)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, MD, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019_Lactose_microbiota
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Bacterial Vaginoses
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Active and inactive tablets were identical. The tablets were packed and labelled by the manufacturer. The key to identity was retained and was disclosed after recruiting all patients. After informed consent, eligible patients drew a closed opaque envelope from a set of envelopes numbered 1-40 and placed in random order. The envelope contained both number labels for medical data-related documents and sample vials and a closed opaque container holding tablets labelled with the sample number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactose (Experimental): Lactose monohydrate 810 mg, silicon dioxide 20 mg, and magnesium stearate 14 mg
  Interventions: Dietary Supplement: Lactose
- Placebo (Placebo Comparator): Dextran 40 EP 671 mg, silicon dioxide 20 mg and magnesium stearate 14 mg
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactose — Lactose monohydrate 810 mg, silicon dioxide 20 mg, and magnesium stearate 14 mg
  Arms: Lactose
Dietary Supplement: Placebo — Dextran 40 EP 671 mg, silicon dioxide 20 mg and magnesium stearate 14 mg
  Arms: Placebo

SUMMARY:
The aim of the study was to investigate whether the administration of a vaginal tablet containing lactose can modulate the bacterial flora of women with bacterial vaginosis (BV).

Design: Double-blind, placebo-controlled randomised trial.

Setting: Women with BV who responded to advertisements in local newspapers and on posters at the Institutions for Education in Health Science in Eastern Jutland, Denmark. These individuals were supplemented with patients enrolled at a gynaecological clinic.

Participants: Forty women with BV diagnosed through the Amsel test. By randomisation, 20 were assigned to receive lactose tablets, and 20 were assigned to receive placebo tablets.

Interventions: Twice daily application of one lactose tablet or placebo tablet for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Amsel criteria positive defined as 3/4 of the following: Vaginal discharge, Fishy odor, pH>4.5 and Clue cells in a wet smear.

Exclusion Criteria:

* Not able to provide written informed consent.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-01 (Actual)

PRIMARY OUTCOMES:
Bacterial load after intervention | 7 days
  quantitative measurements with qPCR for G. vaginalis, Prevotella spp., A. vaginae, Megasphaera type 1, L. gasseri, L. crispatus, L. jensenii and L. iners after intervention